CLINICAL TRIAL: NCT01132677
Title: A Randomized Clinical Trial Comparing Hyaluronic Acid (Hylan G-F 20) and Corticosteroid (Methylprednisolone Acetate) for Knee Osteoarthritis
Brief Title: A Study Comparing Viscosupplementation and Corticosteroid Injections for Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: LifeMark Health (Other)
Responsible Party: Dr. Brad Monteleone, LifeMark Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HA-CS-OA1
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-02

CONDITIONS: Osteoarthritis, Knee
Keywords: OA of Knee; Osteoarthritis of Knee; Viscosupplementation and Osteoarthritis; Viscosupplementation and OA; Hyaluronic Acid; Corticosteroid injection versus hyaluronic acid; Synvisc One and Knee OA; viscosupplementation and knee pain; knee Pain from OA
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Methylprednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronic Acid (HA) Injection (Active Comparator): Patients allocated to the HA group will receive a single IA injection Hylan G-F 20 Synvisc One™ (1 injection of 6cc's). All injections will be administered as outlined on the company label. Aspiration of the knee will not be performed.
  Interventions: Device: Hylan G-F 20 (Synvisc One)
- Corticosteroid Injection (Active Comparator): Patients allocated to the corticosteroid injection will receive a single IA injection of 80mg of methylprednisolone acetate (1cc of solution) mixed with 5cc's of 1% lidocaine without epinephrine for a total of 6cc's. The injection will be administered as outlined on the company label. Aspiration of the knee will not be performed.
  Interventions: Drug: Methylprednisolone (Corticosteroid)

INTERVENTIONS:
Device: Hylan G-F 20 (Synvisc One) — Single IA injection of 6cc's. Injections will be administered as outlined on the company label.
  Arms: Hyaluronic Acid (HA) Injection
Drug: Methylprednisolone (Corticosteroid) — Single IA injection of 80mg of methylprednisolone acetate (1cc of solution) mixed with 5cc's of 1% lidocaine without epinephrine for a total of 6cc's. The injection will be administered as outlined on the company label.
  Arms: Corticosteroid Injection

SUMMARY:
Do differences exist between patients who receive a single intra-articular injection of corticosteroid versus patients who receive a single intra-articular injection of hyaluronic acid for the treatment of knee osteoarthritis at 1, 3 and 6 weeks, and 3 and 6 months post injection?

DETAILED DESCRIPTION:
OBJECTIVES

Primary i. To determine if patients' VAS "pain while walking" is different at 6 weeks post-injection in patients who receive a single injection of methylprednisolone acetate (MPA) versus patients who receive a single injection of Hylan G-F 20 (Synvisc One™) for treatment of knee OA.

Secondary i. To determine if differences in VAS "pain while walking" scores exist at 1 and 3 weeks, and 3 and 6 months post injection between MPA and HA patients.

ii. To determine if differences in VAS "pain at rest" scores exist at 1, 3 and 6 weeks and 3 and 6 months post injection between MPA and HA patients.

iii. To determine if differences in VAS "pain with stairs" scores exist at 1, 3 and 6 weeks and 3 and 6 months post injection between MPA and HA patients.

iii. To determine if differences in KOOS questionnaire scores exist at 6 weeks, 3 months and 6 months post injection between MPA and HA patients.

iv. To determine if differences in WOMAC questionnaire scores exist at 6 weeks, 3 months, and 6 months post injection between MPA and HA patients.

v. To determine if differences in adverse events exist at 1, 3 and 6 weeks, and 3, and 6 months post injection between MPA and HA patients.

vi. To track the number of patients who receive additional injections after 3 months following their index injection.

ELIGIBILITY:
Inclusion Criteria:

* Clinical

  * 19-75 years of age (inclusive)
  * Symptomatic OA (1 of the following: pain, stiffness, or swelling)
  * Evidence of grade I, II or III OA on radiographic images according to Kellgren-Lawrence grading scale.

Exclusion Criteria:

* Clinical

  * Previous surgery on either knee (not including a diagnostic arthroscopy arthroscopy or simple partial meniscectomy)
  * Intra-articular treatment within the last 3 months
  * Ipsilateral cruciate or collateral ligament injury within past 3 months, or evidence of ligament laxity
  * Inflamed knee or pronounced effusion
  * Allergy to birds, eggs, avian proteins or known HA or corticosteroid
  * Venous or lymphatic stasis
  * Skin condition in the injection area
  * Evidence of infection in the affected joint
  * History of crystalline arthropathy or inflammatory arthritis
  * Pregnant or nursing
  * Third Party, Medical Legal or Workers' Compensation Board
  * Patient unable to understand English or unable to providing informed consent

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be "pain while walking for approximately 30 minutes on a flat surface today" as reported by the patient on a 100mm unmarked VAS (0 = no pain; 100 = worst pain possible). | VAS Form will be given at baseline (prior to injection) and then at 1, 3 and 6 weeks, and 3 and 6 months post injection.
  As described in title

SECONDARY OUTCOMES:
Pain at rest or with stairs as reported byu the patient on a VAS | Baseline (pre-injection), 1, 3 and 6 weeks, and 3 and 6 months post injection
  Secondary Outcomes:
  i. "Pain at rest" and "pain with stairs" as reported by the patient on a VAS
  (Additional outcomes ii. Knee injury and Osteoarthritis Outcome Score (KOOS). The KOOS is a valid, reliable and responsive questionnaire that is self-administered and consists of 5 subscales.
  iii. The KOOS includes the WOMAC Osteoarthritis Index LK 3.0 and thus, WOMAC scores will also be computed.
  iv. Adverse events as reviewed and documented by the physician v. The number of subsequent re-injections or treatment strategies.)

CONTACTS AND LOCATIONS:
Overall Officials: Brad J Monteleone, Physician, Principal Investigator — UBC - Department of Family Practice
Locations (1):
- LifeMark Health, Kelowna, British Columbia, Canada